CLINICAL TRIAL: NCT06711107
Title: Predicting Failure of Non-operative Management of Adhesive Small Bowel Obstruction Through Deep Learning.
Brief Title: Predicting NOM Failure in Bowel Obstruction
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Chirdig01
Record Dates: First submitted 2024-11-18; First posted 2024-12-02 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Small Bowel Obstruction; Intestinal Pseudo-Obstruction
MeSH Terms: conditions — Intestinal Pseudo-Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SBO patients: "After adhesive SBO diagnosis is performed through clinical examination, blood tests, and abdominal CT-scan, and need for urgent surgical exploration excluded, patients are admitted to the General/Digestive Surgery Department for NOM. NOM consists in fasting, analgesics, antiemetics, and fluids administration, with or without electrolytes correction. Nasogastric tube positioning and/or hyperosmolar water-soluble contrast administration is not deemed necessary for the patient to be included in this study, thus allowing us to evaluate different management strategies for adhesive SBO.
  After at least 24 hours of NOM, patients are re-evaluated for NOM prosecution or surgical treatment.
  NOM is considered effective when patients achieved symptoms remission, flatus and stools evacuation, and realimentation without symptoms recurrence for at least 90 days.
  NOM failure is defined as need for surgery, both laparoscopic or laparotomic, to treat adhesive SBO. Surgical management depends on single

SUMMARY:
"This study aims to collect data on patients with small bowel obstruction (SBO) admitted to hospitals in France and Italy from May 2022 to October 2024 to develop a deep convolutional neural network (DCNN) model. This model will analyze anonymized CT scans to assess the effectiveness of non-operative management (NOM) for SBO, supporting decisions on surgical intervention. Eligible patients are those diagnosed with SBO due to abdominal adhesions who initially received NOM for at least 24 hours. Patients with other SBO causes, early surgery within 24 hours, or those without a CT scan diagnosis are excluded.

Data collection spans hospitals in Antibes, Nice, Milan, and Vimercate, targeting consecutive SBO cases with adhesive etiology. To perform an external validation of the DCNN, data will also be retrospectively collected from patients admitted to the Antibes hospital between May 2021 and April 2022 with adhesive SBO. This validation set includes patients who underwent NOM successfully and those who needed surgery after NOM failure. The DCNN model will be applied to anonymized, non-contrast and contrast-enhanced portal-phase CT scans of these patients, with researchers blinded to each patient's NOM outcome to prevent bias. The model's performance will then be evaluated using accuracy metrics consistent with those used in initial model testing, ensuring the reliability of results when applied to external cases.

NOM, after adhesive SBO diagnosis via clinical exams, blood tests, and CT scans, includes fasting, analgesics, antiemetics, and fluids as per current guidelines, without necessarily using nasogastric tubes or contrast agents. Patients are re-evaluated after 24 hours to determine whether NOM should continue or if surgery is necessary. NOM is deemed effective if patients experience symptom resolution, stool passage, and no recurrence within 90 days. NOM failure is defined by the need for laparoscopic or laparotomic surgery, based on symptoms' persistence, worsening, or radiological indicators of blockage despite adequate NOM.

Data collection, registered with the French National Committee for Data Protection, includes variables like age, sex, medical history, symptoms, blood tests, CT-scan findings, NOM details, and surgical information. Radiological data, including Digital Imaging and Communication in Medicine (DICOM) files of CT scans, will be anonymized and converted to the Neuroimaging Informatics Technology Initiative (NIfTI) format for secure storage and analysis.

The NIfTI data files will be randomly split into training and test datasets in an 80%-20% ratio, processed separately for non-contrast and contrast-enhanced CT scans. Data augmentation, including random rotation, flipping, zooming, translation, and noise addition, will be applied to improve model accuracy and reduce overfitting. Different DCNN models will be trained and tested and furtherly undergo external validation to produce a tool capable of predicting NOM failure and need for surgery in patients with adhesive SBO."

ELIGIBILITY:
Inclusion Criteria:

* SBO diagnosed through clinical evaluation, blood tests, and an abdominal CT-scan performed at the admission in the Emergency Department.
* SBO secondary to single or multiple abdominal adhesions.
* Initial treatment of SBO by NOM for at least 24 hours.
* Non-opposition to the anonymous data processing by the included patients."

Exclusion Criteria:

* admission for SBO other than of adhesive etiology (hernias, bowel or other abdominal neoplasms, foreign bodies, functional obstruction, etc.).
* surgical treatment of SBO within 24 hours from admission or rather NOM duration < 24 hours.
* SBO diagnosis performed without CT-scan."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The team will collect data from consecutive patients admitted to the Digestive Surgery Department of the Hospital of Antibes (Centre Hospitalier d'Antibes Juan-les-Pins, France) from May the 1st 2022 to October the 31st 2024, to the Digestive and Emergency Surgery Department (Nice University Hospital , France) from the 1st of May 2022 to the 31st of October 2024 , to the General Surgery and Trauma Center of the University Hospital Niguarda in Milan (Grande Ospedale Metropolitano Niguarda, Italy) from the 1st of May 2023 and the 31st of October 2024, and to the General Surgery Department of the Vimercate Hospital (Ospedale di Vimercate, Italy) from the 1st of May 2023 and the 31st of October 2024 with the diagnosis of SBO. Moreover, to perform external validation of the DCNN model, the team will collect data of patients admitted to the Digestive Surgery Department of the Antibes Juan-les-Pins hospital from the 1st of May 2021 to the 30th of April 20
Sampling Method: Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Performance of Deep Learning model in predicting NOM failure | 90 days from patients hospital discharge.
  To measure the degree of agreement between the prediction made by the Deep Learning model and the actual success or failure of non-operative management for small bowel obstruction in the real situation. This will be measured through Area Under the Receiver Operator Characteristic curve (AUROC) assesment. AUROC varies between 0.5 and 1, corresponding to no class separation capacity and full class separation capacity, respectively.

SECONDARY OUTCOMES:
Performance evaluation: accuracy | 90 days from patients hospital discharge.
  The number of true positives and true negatives among all predictions. It varies between 0 (no correct prediction) to 1 (full correct predictions).
Performance evaluation: precision | 90 days from patients hospital discharge.
  The number of true positives divided by all the positive predictions (true positives and false positives). It varies between 0 (no correct prediction) to 1 (full correct predictions)
Performance evaluation: recall | 90 days from patients hospital discharge.
  The number of true positives divided by the actual positive instances in the dataset (true positives and false negatives). It varies between 0 (no correct prediction) to 1 (full correct predictions).
Performance evaluation : balanced accuracy | 90 days from patients hospital discharge.
  the aritmethic mean of sensitivity and specificity. It varies between 0 (no correct prediction) to 1 (full correct predictions).
Performance evaluation:F1-score | 90 days from patients hospital discharge.
  It combines precision and recall. It ranges from 0-100%, and a higher F1 score denotes a better quality classifier.
Performance evaluation: Confusion matrix | 90 days from patients hospital discharge.
  A visual representation of true positives, false positives, true negatives, and false negatives. It is depicted through a table.
Performance evaluation :Log-loss | 90 days from patients hospital discharge.
  It indicates how close the prediction probability is to the corresponding actual/true value (0 or 1 in case of binary classification). The more the predicted probability diverges from the actual value, the higher is the log-loss value.
Performance evaluation: Cohen's Kappa | 90 days from patients hospital discharge.
  A metric used to measure the level of agreement between two raters which can be a useful tool to gauge the performance of a classification model. It accounts for the fact that the raters may happen to agree on some items purely by chance. It varies between 0 (no correct prediction) to 1 (full correct predictions).

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea CHIERICI, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided